CLINICAL TRIAL: NCT04922008
Title: An Open-label, Phase II Study Evaluating the Efficacy and Safety of Trastuzumab Combined With Oral Chemotherapy in Patients With HER-2 Positive Stage I Breast Cancer
Brief Title: Stage I HER2 Positive Invasive Breast Cancer De-escalation Study(IRIS-C/D)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N034
Record Dates: First submitted 2021-06-07; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IRIS-C (Experimental)
  Interventions: Drug: capecitabine and trastuzumab
- IRIS-D (Experimental)
  Interventions: Drug: vinorelbine and trastuzumab

INTERVENTIONS:
Drug: capecitabine and trastuzumab — In IRIS-C cohort, patients who met the inclusion criteria(ER and PR<10%, T≤2cm or ER and/or PR ≥10% 1cm<T≤2cm) would be given capecitabine for 4 cycles with standard trastuzumab for 1 year, in which HR+ patients would be given endocrine therapy for 5 years.
  Arms: IRIS-C
Drug: vinorelbine and trastuzumab — In IRIS-4 cohort, patients who met the inclusion criteria(ER and PR<10%, T≤2cm or ER and/or PR ≥10% 1cm<T≤2cm) would be given vinorelbine for 4 cycles with standard trastuzumab for 1 year, in which HR+ patients would be given endocrine therapy for 5 years.
  Arms: IRIS-D

SUMMARY:
This is an open label, phase II study evaluating the efficacy and safety of trastuzumab combined with oral chemotherapy (capecitabine or vinorelbine) in patients with HER-2 positive stage I breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-70 years old;
* Pathological confirmed of stage I breast cancer: histologically confirmed that the longest diameter of invasive cancer is no more than 2cm and the lymph node is negative (N0);
* If a patient is HR negative(ER/PR<10%), the longest diameter of invasive cancer could not exceed 2cm; while if a patient is HR positive(ER and/or PR ≥10%）,the longest diameter of invasive cancer is greater than 1cm and no more than 2cm;
* The pathological type of immunohistochemistry must meet the following conditions: HER-2 (3+) or HER-2 (0-2 +) with FISH detection is amplified;
* For patients with invasive lesions on both sides, if both lesions are HER-2 positive and meet the tumor size requirements, then can be enrolled;
* Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST)

  ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN#and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula);
* LVEF>50%;
* The patient voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

* Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy;
* Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ;
* Has metastic (Stage 4) breast cancer;
* Pregnant or breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
* Patients participating in other clinical trials at the same time;
* Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmHg, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
* Has severe or uncontrolled infection;
* Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
* The researchers considered patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
iDFS | 5 years
  iDFS invasive disease-free survival

SECONDARY OUTCOMES:
DDFS | 5 years
  distant disease-free survival
OS | 5 years
  overall survival